CLINICAL TRIAL: NCT00001639
Title: Evaluation of Patients With Unresolved Chromosome Aberrations
Brief Title: Evaluation of Patients With Unresolved Chromosome Abnormalities
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970045; 97-HG-0045
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 1999-10

CONDITIONS: Abnormalities; Failure to Thrive; Mental Retardation; Microcephaly
Keywords: Gene Dosage; Haploinsufficiency; Karyotype; Malformations; Mental Retardation
MeSH Terms: conditions — Congenital Abnormalities; Failure to Thrive; Intellectual Disability; Microcephaly

SUMMARY:
The purpose of this research is to study a new way to test for chromosome abnormalities. Chromosomes are strands of DNA (the genetic material in the cell nucleus) that are made up of genes-the units of heredity. Chromosome abnormalities are usually investigated by staining the chromosomes with a dye (Giemsa stain) and examining them under a microscope. This method can detect many duplications and deletions of pieces of chromosomes and is very accurate in diagnosing certain abnormalities. It is not useful, however, for identifying very small abnormalities. This study will evaluate the accuracy of a test method using 24 different dyes for finding small chromosome abnormalities.

Children and adults with various chromosome abnormalities may be eligible for this study, including, for example, people with developmental delay or mental retardation, abnormal growth features or growth retardation, and certain behavioral disorders. Participants will be evaluated in the clinic over a 1- to 3-day period, depending on their symptoms. All participants will be examined by a genetics specialist and will have a physical examination and possibly X-rays, computerized tomography (CT) scans, magnetic resonance imaging (MRI), ultrasound studies and medical photography. Blood will be drawn for chromosome testing-about 3 tablespoons from adults and 1 to 3 teaspoons from children.

When the test results are available, participants will return to the clinic for follow-up evaluation and review of the test findings. The genetic and medical evaluations, along with their implications, will be discussed.

DETAILED DESCRIPTION:
There is a range of genomic aberrations from aneuploidy down to single base pair deletions or inserts. Present technology uses microscopic cytogenetics for detection of large rearrangements (greater than 2 Mb) and molecular techniques for small rearrangements (less than 2 Mb). There is a gap in practical diagnostic technology in that microscopic cytogenetics has poor sensitivity for aberrations less than 5 Mb and the molecular techniques are cumbersome for clinical use in the megabase range. In many cases it is possible to determine that an aberration is present by microscopic cytogenetics but cannot be characterized. We propose to use Spectral Karyotyping (SKY) and supplementary FISH and molecular techniques to characterize these aberrations. Subjects will be seen in OP9 for a clinical genetics evaluation and phlebotomy for SKY. Confirmation of SKY results will be performed by standard FISH, genomic content mapping, and other standard techniques.

ELIGIBILITY:
Physical anomalies or developmental anomalies.

Karyotype showing derivative chromosome abnormality that is not fully characterized.

No abnormal parental karyotype.

No prenatal specimens.

Probands of all ages, genders, and ethnic origin are eligible.

The proband must have a non-mosaic abnormal G-banded chromosome analysis of good quality that shows one or more derivative chromosomes whose foreign component cannot be determined by standard G-banding techniques.

The parents should also have G-banded chromosome analysis prior to eligibility for consent 2. If this has not been done by the referring physician, it may be done as part of the protocol.

The proband with the abnormal karyotype should have one or more of the following features: dysmorphic features; developmental delay or mental retardation; growth retardation, microephaly, short stature or failure to thrive; behavioral disorder

Biological parents must be willing to supply a blood specimen. If they have any of the features listed above, they must attend the clinic if the proband is to be eligible.

The proband must be evaluated by the NCHGR clinical genetics service by the PI, a co-investigator, or his associates.

Mothers will be queried about potential non-paternity. If non-paternity is possible, the family will need to undergo clinical paternity evaluation before they are enrolled in the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 263
Dates: Start 1996-12; Study Completion 2000-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Human Genome Research Institute (NHGRI), Bethesda, Maryland, United States